CLINICAL TRIAL: NCT04677569
Title: ENCORE - A Randomized, Double-Blind, Placebo-Controlled, Active Comparator, Multicenter Study to Evaluate the Efficacy and Safety of an Amikacin Liposome Inhalation Suspension (ALIS)-Based Regimen in Adult Subjects With Newly Diagnosed Nontuberculous Mycobacterial (NTM) Lung Infection Caused by Mycobacterium Avium Complex (MAC)
Brief Title: Study to Evaluate ALIS (Amikacin Liposome Inhalation Suspension) in Participants With Nontuberculous Mycobacterial Lung Infection Caused by Mycobacterium Avium Complex
Acronym: ENCORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS-416; 2020-003079-16 (EudraCT Number); 2023-505273-33-00 (Other: EU CT Number)
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Mycobacterium Infections, Nontuberculous
Keywords: Nontuberculous Mycobacterial Lung Infection; Mycobacterium avium complex; Arikayce®
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous; Mycobacterium avium-intracellulare Infection | interventions — Azithromycin; Ethambutol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALIS + Background Regimen (Experimental): Participants will be administered 590 mg of ALIS (amikacin liposome inhalation suspension) once daily. Participants will also be administered azithromycin 250 mg and ethambutol 15 mg/kg, once daily.
  Interventions: Drug: ALIS; Drug: Azithromycin; Drug: Ethambutol
- ELC + Background Regimen (Placebo Comparator): Participants will be administered ELC (empty liposome control), a visually matching placebo to ALIS (amikacin liposome inhalation suspension), once daily. Participants will also be administered azithromycin 250 mg and ETH (ethambutol) 15 mg/kg, once daily.
  Interventions: Drug: Azithromycin; Drug: Ethambutol; Drug: ELC (matching placebo for ALIS)

INTERVENTIONS:
Drug: ALIS — Inhalation via nebulization over approximately 6 to 15 minutes
  Other Names: Amikacin liposome inhalation suspension; ARIKAYCE®
  Arms: ALIS + Background Regimen
Drug: Azithromycin — Oral tablet
  Other Names: AZI; Zithromax
Drug: Ethambutol — Oral tablet
  Other Names: ETH; Myambutol
Drug: ELC (matching placebo for ALIS) — Inhalation via nebulization over approximately 6 to 15 minutes
  Other Names: Empty liposome control
  Arms: ELC + Background Regimen

SUMMARY:
The main objective of this study is to evaluate the efficacy of ALIS (amikacin liposome inhalation suspension) + background regimen (azithromycin [AZI] + ethambutol [ETH]) compared to the ELC (empty liposome control) + background regimen on participant-reported respiratory symptoms at Month 13.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age (19 years or older in South Korea, 20 years or older in Japan).
* Current diagnosis of MAC lung infection. MAC or mixed infection with MAC as the dominant species is allowed, with MAC as the intended organism for treatment.
* A chest computerized tomography (CT) scan, read locally, within 6 months prior to Screening to determine presence and size of pulmonary cavities. Participants who do not have a chest CT scan within 6 months prior to Screening will be required to obtain a chest CT scan, read locally, during Screening.
* Willingness and ability to adhere to prescribed study treatment during the study.
* Women of childbearing potential (WOCBP) (ie, fertile following menarche and until becoming postmenopausal unless permanently sterile) and fertile men (ie, all men after puberty unless permanently sterile by bilateral orchidectomy) agree to practice a highly effective method of birth control from Day 1 to at least 90 days after the last dose. Examples of such birth controls are:

  * true abstinence (refraining from heterosexual intercourse during the entire study),
  * copper intrauterine device (IUD),
  * hormonal methods (levonorgestrel-releasing intrauterine system, progestogen implant, combined oral contraceptive pill [combined with barrier method]),
  * exclusive homosexual relationship, or
  * sole male partner who has undergone surgical sterilization with confirmation of azoospermia at least 3 months post procedure.
* Provide signed informed consent prior to administration of study drugs or performing any study-related procedure.
* Be able to comply with study drugs use, study visits, and study procedures as defined by the protocol.
* Men with partners who are WOCBP (pregnant or non-pregnant) agree to use condoms and non-pregnant partners should practice a highly effective method of birth control

Exclusion Criteria:

* Diagnosis of cystic fibrosis (CF).
* History of more than 3 MAC lung infections (a 4th MAC lung infection is not eligible)
* Received any mycobacterial antibiotic treatment for current MAC lung infection
* Refractory MAC lung infection, defined as having positive MAC cultures while being treated with a multidrug mycobacterial antibiotic treatment regimen for a minimum of 6 consecutive months and no documented successful treatment, defined as negative sputum culture for MAC and cessation of treatment
* Relapse of prior MAC lung infection, defined as positive sputum culture for MAC ≤6 months of cessation of prior successful treatment
* Evidence of any pulmonary cavity ≥ 2 cm in diameter, as determined by chest CT scan, read locally, during Screening or within 6 months prior to Screening
* Radiographic finding of new lobar consolidation, atelectasis, significant pleural effusion, or pneumothorax during routine clinical care within 2 months prior to Screening
* Active pulmonary malignancy (primary or metastatic) or any malignancy requiring chemotherapy or radiation therapy within 1 year prior to Screening or anticipated during the study
* Acute pulmonary exacerbation (eg, chronic obstructive pulmonary disease (COPD) or bronchiectasis) requiring treatment with antibiotics, or corticosteroids (intravenous [IV] or oral), within 4 weeks prior to and during Screening
* Current smoker
* History of lung transplantation
* Prior exposure to ALIS (including clinical study)
* Known hypersensitivity or contraindications to use to ALIS, aminoglycosides, or any of their excipients
* Disseminated MAC infection
* Administration of any investigational drug within 8 weeks prior to Screening
* Known or suspected acquired immunodeficiency syndromes (Human Immunodeficiency Virus (HIV) -positive, regardless of CD4 counts). Other immunodeficiency syndromes that may interfere with study participation in the opinion of the Investigator
* Current alcohol, medication, or illicit drug abuse
* Known and active COVID-19 infection
* Known hypersensitivity or contraindications to use of ethambutol, azithromycin (including other macrolides or ketolides), or any of their excipients per local labeling guidance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Respiratory Symptom Score at Month 13 | Baseline to Month 13

SECONDARY OUTCOMES:
Percentage of Participants Achieving Durable Culture Conversion at Month 15 | Month 15
Change from Baseline in Fatigue Symptom Score at Month 13 | Baseline to Month 13
Percentage of Participants Achieving Culture Conversion by Month 6 | Month 6
Percentage of Participants Achieving Culture Conversion by Month 12 | Month 12
Percentage of Participants Achieving Culture Conversion by Month 13 | Month 13
Percentage of Participants Achieving Culture Conversion During Treatment | Baseline to Month 12
Time to Culture Conversion | Baseline to Month 12
Time to the First Negative Culture | Baseline to Month 12
Percentage of Participants Who Develop a Mycobacterium avium Complex (MAC) Isolate with Amikacin Minimum Inhibitory Concentration (MIC) ≥ 128 μg/mL More Than One Time | Baseline to Month 15
Percentage of Participants Achieving Culture Conversion and a Subsequent at Least one MAC Positive Culture in Agar Media or Broth Media in at Least 2 Consecutive Visits With Matching Species and Genome at Screening/ Baseline | Baseline to Month 15
Percentage of Participants Achieving Culture Conversion and a Subsequently have at least One MAC Positive Culture in Agar Media or Broth Media in at Least 2 Consecutive Visits With Differing Species and/or Genome at Screening/ Baseline | Baseline to Month 15
Percentage of Participants Meeting the Within-subject Meaningful Change Threshold as Reflected in the Change in Respiratory Symptom Scores Computed From Baseline to Month 13 | Baseline to Month 13
Number of Participants Who Experience an Adverse Event (AEs) | Baseline to Month 15

CONTACTS AND LOCATIONS:
Locations (258):
- United States (90):
  - USA008, Birmingham, Alabama
  - USA062, Fresno, California
  - USA060, Los Angeles, California
  - USA090, Newport Beach, California
  - USA058, Sacramento, California
  - USA048, San Diego, California
  - USA081, San Francisco, California
  - USA055, Santa Barbara, California
  - USA050, Stanford, California
  - USA001, Denver, Colorado
  - USA023, Washington D.C., District of Columbia
  - USA080, Bradenton, Florida
  - USA028, Brandon, Florida
  - USA003, Clearwater, Florida
  - USA043, Jacksonville, Florida
  - USA072, Jacksonville, Florida
  - USA085, Jacksonville, Florida
  - USA047, Jacksonville, Florida
  - USA042, Kissimmee, Florida
  - USA019, Leesburg, Florida
  - USA039, Naples, Florida
  - USA096, Naples, Florida
  - USA097, Naples, Florida
  - USA046, New Port Richey, Florida
  - USA054, Sarasota, Florida
  - USA084, Sebastian, Florida
  - USA026, Sebring, Florida
  - USA070, St. Petersburg, Florida
  - USA014, St. Petersburg, Florida
  - USA067, Tampa, Florida
  - USA068, Tampa, Florida
  - USA053, Weston, Florida
  - USA038, Atlanta, Georgia
  - USA066, Augusta, Georgia
  - USA004, Lawrenceville, Georgia
  - USA029, Rincon, Georgia
  - USA079, Coeur d'Alene, Idaho
  - USA031, Chicago, Illinois
  - USA073, Springfield, Illinois
  - USA030, Springfield, Illinois
  - USA074, Iowa City, Iowa
  - USA037, Kansas City, Kansas
  - USA002, New Orleans, Louisiana
  - USA017, Baltimore, Maryland
  - USA099, Lexington, Massachusetts
  - USA077, Springfield, Massachusetts
  - USA013, Rochester, Minnesota
  - USA082, Columbia, Missouri
  - USA061, St Louis, Missouri
  - USA045, Omaha, Nebraska
  - USA009, Omaha, Nebraska
  - USA069, Hillsborough, New Jersey
  - USA032, Toms River, New Jersey
  - USA065, Bayside, New York
  - USA088, East Syracuse, New York
  - USA011, New York, New York
  - USA059, The Bronx, New York
  - USA076, Charlotte, North Carolina
  - USA035, Charlotte, North Carolina
  - USA033, Charlotte, North Carolina
  - USA051, Durham, North Carolina
  - USA034, Mooresville, North Carolina
  - USA007, Winston-Salem, North Carolina
  - USA075, Cincinnati, Ohio
  - USA064, Cincinnati, Ohio
  - USA018, Cleveland, Ohio
  - USA063, Columbus, Ohio
  - USA071, Portland, Oregon
  - USA025, Portland, Oregon
  - USA015, DuBois, Pennsylvania
  - USA040, Philadelphia, Pennsylvania
  - USA093, Philadelphia, Pennsylvania
  - USA092, Providence, Rhode Island
  - USA044, Anderson, South Carolina
  - USA024, Charleston, South Carolina
  - USA020, Charleston, South Carolina
  - USA012, Rock Hill, South Carolina
  - USA022, Franklin, Tennessee
  - USA041, Hendersonville, Tennessee
  - USA078, Nashville, Tennessee
  - USA016, Dallas, Texas
  - USA100, Dallas, Texas
  - USA091, Denison, Texas
  - USA086, Houston, Texas
  - USA021, McKinney, Texas
  - USA006, San Antonio, Texas
  - USA089, Temple, Texas
  - USA052, Tyler, Texas
  - USA083, Charlottesville, Virginia
  - USA087, Madison, Wisconsin
- Argentina (7):
  - ARG004, Ciudad autAnoma de Buenos Aires, Buenos Aires
  - ARG005, Quilmes, Buenos Aires
  - ARG006, Villa Vatteone, Buenos Aires
  - ARG003, CArdoba, CArdoba
  - ARG002, Córdoba, CArdoba
  - ARG001, Rosario, Santa Fe Province
  - ARG007, San Miguel de Tucumán, Tucumán Province
- Australia (16):
  - AUS006, Concord, New South Wales
  - AUS004, New Lambton Heights, New South Wales
  - AUS002, Westmead, New South Wales
  - AUS012, Birtinya, Queensland
  - AUS010, Chermside, Queensland
  - AUS013, Douglas, Queensland
  - AUS003, Greenslopes, Queensland
  - AUS016, Herston, Queensland
  - AUS014, Meadowbrook, Queensland
  - AUS001, South Brisbane, Queensland
  - AUS011, Woolloongabba, Queensland
  - AUS008, Adelaide, South Australia
  - AUS007, Clayton, Victoria
  - AUS009, Melbourne, Victoria
  - AUS015, Spearwood, Western Australia
  - AUS005, Perth
- Austria (2):
  - AUT003, Wels, OberAsterreich
  - AUT001, Linz, Upper Austria
- Belgium (3):
  - BEL003, Brussels, Brussels Capital
  - BEL002, Ghent
  - BEL001, Leuven
- Canada (3):
  - CAN003, Winnepeg, Manitoba
  - CAN002, Toronto, Ontario
  - CAN004, Windsor, Ontario
- Chile (4):
  - CHL001, Curicó, Maule Region
  - CHL002, Quillota
  - CHL004, Talca
  - CHL003, Valparaíso
- Denmark (5):
  - DNK005, Vejle, Region Syddanmark
  - DNK001, Roskilde, Zeeland
  - DNK004, Aalborg
  - DNK002, Aarhus N
  - DNK003, Odensa C
- France (16):
  - FRA012, Nice, Alpes-Maritimes
  - FRA016, Strasbourg, Bas-Rhin
  - FRA015, Pessac, Gironde
  - FRA010, Suresnes, Hauts-de-Seine
  - FRA008, Nantes, Loire-Atlantique
  - FRA006, Amiens
  - FRA005, Brest
  - FRA007, Caen
  - FRA002, Créteil
  - FRA001, Marseille
  - FRA014, Paris
  - FRA009, Paris
  - FRA013, Paris
  - FRA004, Saint-Denis
  - FRA003, Saint-Pierre
  - FRA011, Toulouse
- Germany (14):
  - GER001, Donaustauf, Bavaria
  - GER013, Gauting, Bavaria
  - GER005, München, Bavaria
  - GER012, Potsdam, Brandenburg
  - GER010, Immenhausen, Hesse
  - GER003, Borstel, Lower Saxony
  - GER014, Cologne, North Rhine-Westphalia
  - GER011, Cologne, North Rhine-Westphalia
  - GER008, Berlin
  - GER006, Dresden
  - GER009, Essen
  - GER002, Frankfurt
  - GER004, Freiburg im Breisgau
  - GER007, Hanover
- Greece (3):
  - GRC002, Athens, Attica
  - GRC003, Alexandroupoli
  - GRC001, Heraklion
- Hungary (2):
  - HUN002, Budapest
  - HUN001, Törökbálint
- Israel (7):
  - ISR008, Tel Aviv, Tel Aviv
  - ISR001, Ashkelon
  - ISR002, Beer-Yaakov
  - ISR007, Haifa
  - ISR005, Jerusalem
  - ISR003, Petah Tikva
  - ISR004, Ramat Gan
- Italy (11):
  - ITA006, Modena, Emilia-Romagna
  - ITA011, Reggio Emilia, Emilia-Romagna
  - ITA010, Genoa, Liguria
  - ITA002, Milan, Milano
  - ITA008, Siena, Tuscany
  - ITA004, Florence
  - ITA001, Milan
  - ITA009, Milan
  - ITA007, Monza
  - ITA003, Pavia
  - ITA005, Roma
- Japan (21):
  - JPN011, Nagoya, Aiti
  - JPN020, Kita Kyushu-shi, Hukuoka
  - JPN022, Yokohama-Shi Tsuzuki-Ku, Kanagawa
  - JPN017, Matsusaka-Shi, Mie-ken
  - JPN018, Nagasaki, Nagasaki
  - JPN023, Kurashiki-Shi, Okayama-ken
  - JPN019, Izumo-Shi, Shimane
  - JPN014, Hamamatsu, Shizuoka
  - JPN015, Kiyose-Shi, Tokyo
  - JPN021, Ōta-ku, Tokyo
  - JPN008, Shinjuku-ku, Tokyo
  - JPN001, Fukui
  - JPN004, Fukuoka
  - JPN003, Jonan-ku
  - JPN010, Kiyose
  - JPN006, Nagano
  - JPN012, Naka-gun
  - JPN002, Sakaishi
  - JPN009, Shimonoseki
  - JPN005, Tokyo
  - JPN016, Toyonaka-Shi, Ôsaka
- New Zealand (4):
  - NZL003, Hastings, Hawkes's Bay
  - NZL002, Hamilton, Waikato Region
  - NZL004, Auckland
  - NZL001, Christchurch
- POL003, Kielce, Świętokrzyskie Voivodeship, Poland
- Portugal (2):
  - PRT002, Braga
  - PRT003, Lisbon
- South Korea (9):
  - KOR008, Ansan-si, Gyeonggido
  - KOR005, Seongnam-si, Gyeonggido
  - KOR007, Seongbuk-Gu, Seoul Teugbyeolsi
  - KOR006, Incheon
  - KOR004, Seoul
  - KOR002, Seoul
  - KOR009, Seoul
  - KOR003, Seoul
  - KOR001, Seoul
- Spain (12):
  - ESP009, L'Hospitalet de Llobregat, Barcelona
  - ESP007, Vigo, Pontevedra
  - ESP002, Barcelona
  - ESP008, Barcelona
  - ESP003, Barcelona
  - ESP005, Girona
  - ESP010, Madrid
  - ESP001, Madrid
  - ESP004, Madrid
  - ESP011, Pamplona
  - ESP006, Pontevedra
  - ESP012, Seville
- Taiwan (12):
  - TWN004, Chiayi City, Chiayi
  - TWN001, Douliu
  - TWN012, Hsinchu
  - TWN005, Kaohsiung City
  - TWN003, Kaohsiung City
  - TWN007, New Taipei City
  - TWN006, Taipei
  - TWN011, Taipei
  - TWN010, Taipei
  - TWN008, Taipei
  - TWN009, Taipei
  - TWN002, Taipei
- Turkey (Türkiye) (3):
  - TUR004, Maltepe, Istanbul
  - TUR003, Izmir
  - TUR002, Kocaeli
- United Kingdom (11):
  - GBR009, Plymouth, Devon
  - GBR012, Salford, Lancashire
  - GBR013, Swansea, West Glamorgan
  - GBR008, Birmingham, West Midlands
  - GBR005, Aberdeen
  - GBR001, Cambridge
  - GBR002, Dundee
  - GBR004, Liverpool
  - GBR007, London
  - GBR010, London
  - GBR003, London

IPD SHARING:
Plan to Share IPD: No